CLINICAL TRIAL: NCT03199144
Title: Neoadjuvant Chemotherapy and Stereotactic Radiosurgery to Pancreatectomy for Borderline Resectable Pancreatic Cancer : Phase II Study
Brief Title: Neoadjuvant Chemotherapy and Stereotactic Radiosurgery to Pancreatectomy for Patients With Borderline Resectable Pancreatic Cancer
Acronym: CKPancreas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties to recruit patients
Sponsor: Centre Francois Baclesse, Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pancreas cancer neoadjuvant
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Neoplasms; Borderline resectable; Neoadjuvant treatment; Chemotherapy; Stereotactic radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic radiotherapy (Experimental): Stereotactic radiotherapy delivering 30 Gy in 5 fractions over 9 days
  Interventions: Drug: Chemotherapy; Radiation: Stereotactic radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Chemotherapy — 3 cycles of Gemzar-Abraxane
Radiation: Stereotactic radiotherapy — Stereotactic radiation treatment delivering 30 Gy in 5 fractions over 9 days
Procedure: Surgery — Whipple procedure will be the recommended procedure but will be modified according to the initial tumor location

SUMMARY:
The goal of the present study is to test if in situations of borderline resectable patients a neoadjuvant treatment combining Gemzar-Abraxane and stereotactic radiosurgery could increase the median OS rates above 30 months that means at least 12 months more than the 18-20 months generally described.

DETAILED DESCRIPTION:
1. Chemotherapy : 3 cycles of Gemzar-Abraxane. Nab-Paclitaxel will be delivered at day 1 at the dose of 125mg/m2. Gemcitabine will be delivered at the dose of 1g/m2 at days 1, 8 and 15. Three cycles will be given at 4 weeks intervals.

2. PET Scanner and Magnetic resonance Imaging within the 10 days of the third chemotherapy cycle

3.Radiation treatment: Stereotactic radiation treatment delivering 30 Gy in 5 fractions over 9 days, according to the ongoing "CYM 6 Spinal CFB1" which was approved by the "Centre National d'Ethique et de Recherches" (CNER) under the Number 20013/1103 (Ongoing Study 3).

At first, 4 coïl fiducials will be placed inside and/or around the tumor. 10 days later the imaging preparation procedure will be initiated with a CT Scan and MRI simulation. Both exams will be fused using the fiducials. The Clinical Target Volume (CTV) will include systematically the coeliac trunk until the aorta with a margin of at least 1 cm, the origin of the upper mesenteric vessels until the aorta with at least a margin of 1 cm, the space between the Inferior Cava Vein (ICV) and the aorta in front of the pancreatic region, the space between the portal vein and ICV and finally the right lateral border of the ICV in front of the pancreatic region in case of pancreatic head tumors only. The CTV will also include the tumor mass with a 1 cm margin and the locally positive CT scan or PET scanner nodes with a margin of 1 cm provided it does not overlay the digestive structures that will remain after the surgical resection. Finally all these regions will be linked to make a unique CTV structure. The PTV will be defined as an expansion of 5 mm from the CTV. The doses tolerated to the organs at risk figure in the Ongoing Study 3.

Radiation treatment will be initiated 4 weeks after the third chemotherapy cycle.

4. Surgery : Whipple procedure will be the recommended procedure but will be modified according to the initial tumor location. The extension degree of the resection will remain at the discretion of the surgeon. However all the bowel and duodenum irradiated at the prescription dose will be systematically removed whatever the importance of the surgical resection.

Minimal Follow up :

1. Clinical exam every 3 months for 3 years
2. Thoraco-abdominal CT scan at 6, 12, 18, 24, 30 and 36months
3. PET Scanner at 6, 12, 18, 24, 30 and 36months
4. CA 19.9 every 3 months for 3 years

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven pancreatic adenocarcinoma
* Borderline resectable pancreatic adenocarcinoma (NCCN guidelines)
* OMS status ≤2
* Age at presentation >18 y
* Absolute neutrophil counts >1500/ml
* Absolute platelet count >100000/ml
* GOT and GPT <2.5 x the upper limit of normal
* Total bilirubin < the upper limit of normal
* Serum creatinin < upper limit of normal
* Coagulation test within limit of normal (Prothrombin time, INR) +/- 15%
* No evidence of jaundice at enrolment. If stent required to alleviate jaundice it should be metallic
* Patient must be able to eat without a feeding tube and can take medications orally
* Disease must be encompassed in a reasonable radiation field
* Signed informed consent

Exclusion Criteria:

* Distant metastases
* Evolutive disease after the neoadjuvant chemotherapy course according RECIST criteria
* Neuroendocrine tumors
* Peritoneal dissemination visualized at diagnostic abdominal CT scan
* Pathologic abdominal nodes visualized at diagnostic abdominal CT scan outside the pancreatic area
* Pathologic PET scan outside the pancreatic area
* Inoperability for medical reasons
* Inability to tolerate chemotherapy for medical (in particular grade II or more neuropathy) or allergic purposes, or for OMS score >2
* Inability to tolerate Whipple resection
* Collagenose diseases
* Cancer evolution outside the pancreatic bed at the PET scanner performed just after the 3 neo adjuvant chemotherapy cycles
* Any previous cancer in the 5 years excepted a basal skin cell carcinoma or in situ cervical cancer
* Active infection with HIV, Hepatitis B or c
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
patient overall survival | follow up during 3 years after patient inclusion
  patient overall survival

SECONDARY OUTCOMES:
positive surgical margins | follow up during 3 years after patient inclusion
  assessment of R1 margin defined according to the British Royal College of pathology
toxicity according the CTCAEv4 | follow up during 3 years after patient inclusion
  toxicity according the CTCAEv4
CA19.9 level post operatively | follow up during 3 years after patient inclusion
  CA19.9 levels post operatively
CEA level post operatively at one month | follow up during 1 month after patient inclusion
  CEA level post operatively at one month

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Esch-sur-Alzette, SUD, Luxembourg

IPD SHARING:
Plan to Share IPD: No